CLINICAL TRIAL: NCT07329582
Title: A Prospective, Double-blinded, Randomised Controlled Trial Comparing the Use of Hyperbaric Bupivacaine Versus Hyperbaric Prilocaine for Spinal Anaesthesia in Asian Patients Undergoing Elective Total Knee Replacement
Brief Title: Hyperbaric Bupivacaine Versus Hyperbaric Prilocaine in Spinal Anaesthesia
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023/00591
Record Dates: First submitted 2025-12-21; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Knee Replacement, Total; Knee Replacement Surgery
Keywords: total knee replacement; spinal anaesthesia; Bupivacaine; Prilocaine
MeSH Terms: interventions — Prilocaine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to receive either prilocaine or bupivacaine for their spinal anesthesia
Who Masked: Participant, Outcomes Assessor
Masking Description: This helps to eliminate potential placebo effects or bias in self-reported outcomes. The masking of outcome assessors ensures that the individuals evaluating the results of the trial are unaware of which treatment each participant received. By masking both participants and outcome assessors, the study aims to minimize bias and increase the reliability of the results, as neither the subjects nor those evaluating their progress can be influenced by knowledge of the treatment assignment."
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bupivacaine (Other): The administration of the spinal anesthetic will follow the hospital's standard protocol for this procedure. This means that apart from the specific local anesthetic used (prilocaine or bupivacaine), all other aspects of the anesthesia process - including patient preparation, sterile technique, needle size and type, patient positioning, and post-procedure care - will remain consistent with the hospital's established guidelines for spinal anesthesia
  Interventions: Drug: prilocaine
- prilocaine (Active Comparator): The administration of the spinal anesthetic will follow the hospital's standard protocol for this procedure. This means that apart from the specific local anesthetic used (prilocaine or bupivacaine), all other aspects of the anesthesia process - including patient preparation, sterile technique, needle size and type, patient positioning, and post-procedure care - will remain consistent with the hospital's established guidelines for spinal anesthesia
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: prilocaine — Prilocaine is known to have a faster recovery time by producing a shorter duration of motor block and less urinary retention, this results in a more rapid rehabilitation in post-total knee replacement surgical patients
  Arms: bupivacaine
Drug: Bupivacaine — Bupivacaine has long been the go-to choice for spinal anesthesia in total knee replacement surgeries due to its effectiveness in providing surgical anesthesia
  Arms: prilocaine

SUMMARY:
Prilocaine numbs you for a shorter time, allowing you to regain movement quicker, which helps you recover faster, start rehab sooner, and feel more satisfied with your treatment overall.

DETAILED DESCRIPTION:
Bupivacaine has long been the go-to choice for spinal anesthesia in total knee replacement surgeries due to its effectiveness in providing surgical anesthesia. However, it comes with some drawbacks, primarily its prolonged motor block and the potential for dose-related hypotension, which can hinder post-operative recovery. In contrast, prilocaine has gained popularity in recent years, particularly for outpatient procedures and even caesarean sections. Prilocaine's appeal lies in its faster recovery profile, characterized by a shorter duration of motor block and reduced incidence of urinary retention. These properties make it an attractive option for total knee replacement patients, as it potentially allows for quicker rehabilitation. The shorter-acting nature of prilocaine means patients may regain mobility sooner, potentially leading to earlier discharge and improved overall satisfaction. Despite these promising attributes, there's a notable gap in research comparing the intrathecal use of hyperbaric prilocaine 2% with hyperbaric bupivacaine 0.5%, especially within the Asian population. This lack of comparative studies highlights the need for further investigation to determine if prilocaine's benefits observed in other contexts translate effectively to total knee replacement procedures in Asian patients, potentially offering a pathway to enhanced recovery protocols in this specific demographic.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective unilateral total knee replacement
* Able to give informed consent

Exclusion Criteria:

* Patients of age < 21 or > 90 years old
* American Society of Anaesthesiologists (ASA) physical status> III
* Extremes of weight: <40kg or BMI >40
* Contra-indications to spinal anaesthesia, prilocaine or bupivacaine (including allergy to local anaesthesia agents or patients at high risk for methaemoglobinemia)
* Complex TKR as deemed by surgeons
* Patient refusal
* Failure of spinal anaesthesia resulting in conversion to general anaesthesia, prior to start of operation
* Patients with prostate hyperplasia or urogenital pathologies
* Planning to conceive / pregnant women / breastfeeding

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Duration of Motor Block | Measured from the time of spinal anesthesia administration until full motor recovery, expected within 24 hours post-operation.
  This study will measure the duration of motor block, defined as the time from spinal anesthesia administration to full recovery of motor function. Motor function will be assessed using the modified Bromage scale, with full recovery defined as a Bromage score of 0 (full movement of legs and feet). The primary hypothesis is that prilocaine will produce an effective sensory block while resulting in a significantly shorter duration of motor block compared to bupivacaine. Assessments will be conducted at regular intervals following the administration of spinal anesthesia until full motor recovery is achieved, with an expected timeframe of up to 24 hours post-operation. This outcome measure will help determine the comparative efficacy of prilocaine versus bupivacaine in facilitating earlier mobilization and potentially enhancing post-operative recovery in patients undergoing total knee replacement surgery.

SECONDARY OUTCOMES:
Comparison of Side Effects between Prilocaine and Bupivacaine | From spinal anesthesia administration up to 24 hours post-operation.
  The study will assess the overall incidence and severity of anesthesia-related adverse events associated with intrathecal prilocaine and bupivacaine in patients undergoing total knee replacement surgery. The measure encompasses a comprehensive range of potential physiological, neurological, and systemic reactions typically associated with spinal anesthesia and local anesthetic use.

CONTACTS AND LOCATIONS:
Overall Officials: Jasmin Jeanette Tan, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No